CLINICAL TRIAL: NCT05670925
Title: The Opportune Administration of Nab-paclitaxel in the First Line Treatment Strategy, Camrelizumab and Famitinib With/Without Nab-paclitaxel, of Patients With Unresectable Locally Advanced or Metastatic Immunomodulatory Triple Negative Breast Cancer：An Open, Single-arm, Multicenter Phase II Clinical Study.
Brief Title: A Trial Exploring the Opportune Administration of Nab-paclitaxel in the First Line Treatment, Camrelizumab Combined With Nab-paclitaxel and Famitinib, of TNBC.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-plus-Pairs
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab plus Famitinib with/without nab-palitaxel (Experimental)
  Interventions: Drug: Camrelizumab plus Famitinib with/without nab-Palitaxel

INTERVENTIONS:
Drug: Camrelizumab plus Famitinib with/without nab-Palitaxel — After enrollment confirmed, the regimen of Camrelizumab Combined with Famitinib will be conducted for 2 cycles (8 weeks). Patients of CR or PR after 2 cycles (8 weeks) will enter dual-therapy maintenance phase until disease progression and will be recorded as PFS-1α. Patients of PD after 2 cycles (8 weeks) will be recorded as PFS-1β. Patients of SD with 2 cycles of dual therapy wlii receive triple therapy regimen: Camrelizumab and Famitinib with nab-Paclitaxel.

SUMMARY:
The study is being conducted to evaluate the Opportune Administration of Nab-paclitaxel in the First Line Treatment Strategy, Camrelizumab and Famitinib with/without Nab-paclitaxel, of Patients with Unresectable Locally Advanced or Metastatic Immunomodulatory Triple Negative Breast Cancer.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status of 0-1
* Expected lifetime of not less than three months
* Metastatic or locally advanced, histologically documented TNBC (absence of HER2, ER, and PR expression)
* Cancer stage: recurrent or metastatic breast cancer; Local recurrence be confirmed by the researchers could not be radical resection.
* Adequate hematologic and end-organ function, laboratory test results.
* Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1) • Patients had received no previous chemotherapy or targeted therapy for metastatic triple-negative breast cancer

Exclusion Criteria:

* Previous received anti-VEGFR small molecule tyrosine kinase inhibitors (e.g. famitinib, sorafenib, Sunitinib, regorafenib, etc.) for treatment of the patients .
* A history of bleeding, any serious bleeding events.
* Important blood vessels around tumors has been infringed and high risk of bleeding.
* Coagulant function abnormality
* artery/venous thromboembolism event
* History of autoimmune disease
* Positive test for human immunodeficiency virus
* Active hepatitis B or hepatitis C
* Uncontrolled pleural effusion and ascites • Known central nervous system (CNS) disease.
* Long-term unhealing wound or incomplete healing of fracture
* urine protein ≥2+ and 24h urine protein quantitative > 1 g.
* Pregnancy or lactation.
* Thyroid dysfunction.
* Peripheral neuropathy grade ≥2.
* People with high blood pressure;
* A history of unstable angina;
* New diagnosis of angina pectoris.
* Myocardial infarction incident ;

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 46 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
PFS | max 24 months
  Progression Free Survival

SECONDARY OUTCOMES:
ORR | 8 WEEKS
  Objective Response Rate according to RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center Shanghai, China, 200032, Shanghai, Shanghai Municipality, China